CLINICAL TRIAL: NCT06769594
Title: Clinical Feasibility and Evaluation of Silicon Photon Counting CT
Brief Title: Next Generation CT System
Status: Recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: SA-000001
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- General: Approximately 80 subjects whose standard of care imaging involved the head/neck, chest, abdomen/bowel and/or musculoskeletal regions will be enrolled.
  Interventions: Device: Investigational CT Scan
- Cardiac: Approximately 20 subjects whose standard of care imaging involved the heart will be enrolled.
  Interventions: Device: Investigational CT Scan

INTERVENTIONS:
Device: Investigational CT Scan — All pre-contrast testing and administration of supporting medications shall be done according to the hospital's SOC. Images will then be compared with the previously acquired imaging conducted as standard of care. The investigational scan takes between 10-30 minutes.

SUMMARY:
The purpose of the study is to collect data to evaluate utility of a next generation CT system in a clinical setting.

DETAILED DESCRIPTION:
Data collected in this study includes an assessment of image quality parameters including spatial resolution, image contrast, and noise to evaluate the product. This data and analysis will help support regulatory submission.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in this study if they meet the following criteria:

1. Who are 18 year of age or older;
2. Able to sign and date the informed consent form; AND
3. Who have in the past 120 days or will in the future 30 days from the day of consent undergo a clinically indicated imaging exam (MRI, CT, radiograph, nuclear medicine, ultrasound, bone material density, interventional radiology procedure) of the head, neck, heart, chest, abdomen, pelvis, or extremities where images are available for this prior exam.

Exclusion Criteria:

Subjects may be excluded from participating in study if they meet any of the following criteria:

1. Who are pregnant or lactating;
2. Who were previously enrolled in this study;
3. For contrast-enhanced CT exams, anyone with known or suspected allergy to iodinated contrast agents;
4. For contrast-enhanced CT exams, anyone with known or suspected renal insufficiency as determined by site medical personnel;
5. Who are in need of urgent or emergent care;
6. Who have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject; and,
7. Who are unwilling to have GEHC personnel present for the CT exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults that are 18-years of age or older, and who have undergone a prior clinically indicated imaging exam of at least one of the following anatomical areas: head, neck, heart, chest, abdomen, pelvis, and/or extremities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 12 months
  Number of investigational CT scans along with standard of care CT images

SECONDARY OUTCOMES:
Safety Information | 12 months
  Type and numbers of AEs, SAEs, and Device Deficiencies
Assessment of Image Quality | 12 months
  Images created from the raw investigational CT scan data will be scored for image quality

CONTACTS AND LOCATIONS:
Overall Officials: MICT Global Research Manager, Study Director — GE Healthcare
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No